CLINICAL TRIAL: NCT02359318
Title: Enamel Damages Following De-bracketing of Demineralised Teeth With or Without Prior Infiltration Compared to Sound Enamel: A Single-center, Randomized, Single Blinded, Split-mouth Controlled Clinical Trial
Brief Title: Enamel Damages Following De-bracketing From Infiltrated Surfaces
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DMG Dental Material Gesellschaft mbH (Industry)
Collaborators: Universidad de La Frontera (Other); Universidad de Concepcion (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RIDeBond
Record Dates: First submitted 2015-01-22; First posted 2015-02-10 (Estimated); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Dental White Spots
Keywords: White spot lesion; Resin Infiltration; Icon; Debonding; Enamel damages; Orthodontic white spots; Orthodontics
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Resin infiltration and de-bonding (Experimental): Patients with brackets and white spots are included in this group. After removal of the old brackets the quadrants are randomized to this intervention arm and the "no infiltration and de-bonding" arm. The teeth that are included in this intervention arm are treated by resin infiltration using Icon (DMG, Germany) according to the manufacturers´ instruction. This is followed by bonding of new brackets (Gemini metal brackets, 3M Unitek). These new brackets are finally de-bonded 4 weeks after the treatment, with silicon impressions taken before adhesive removal.
  Bonding and debonding of brackets is performed by one clinician (Roberto Vogel) using the same bonding and de-bonding techniques and materials for all patients.
  Interventions: Procedure: Resin infiltration; Procedure: Bonding and debonding of brackets.
- No infiltration and de-bonding (Placebo Comparator): Patients with brackets and white spots are included in this group. After removal of the old brackets the quadrants are randomized to this intervention arm and the "resin infiltration and de-bonding" arm. The teeth that are included in this intervention arm are left untreated new brackets (Gemini metal brackets, 3M Unitek) are bonded. These new brackets are finally de-bonded 4 weeks after the treatment, with silicon impressions taken before adhesive removal.
  Bonding and debonding of brackets is performed by one clinician (Roberto Vogel) using the same bonding and de-bonding techniques and materials for all patients.
  Interventions: Procedure: Bonding and debonding of brackets.
- Control and de-bonding (Other): Patients with brackets and without white spots are included in this group. After removal of the old brackets, new brackets (Gemini metal brackets, 3M Unitek) are bonded again. These new brackets are finally de-bonded 4 weeks after the treatment, with silicon impressions taken before adhesive removal.
  Bonding and debonding of brackets is performed by one clinician (Roberto Vogel) using the same bonding and de-bonding techniques and materials for all patients.
  Interventions: Procedure: Bonding and debonding of brackets.

INTERVENTIONS:
Procedure: Resin infiltration — Resin infiltration is done according to manufactures´ instructions after de-bonding of old brackets and prior bonding of new brackets.
  Other Names: Icon (DMG, Germany), Approximal resin infiltration kit
  Arms: Resin infiltration and de-bonding
Procedure: Bonding and debonding of brackets. — Brackets (Gemini metal brackets (3M Unitek) are bonded and de-bonded by one clinician (Roberto Vogel) and using the same bonding and de-bonding techniques and materials for all patients. All brackets were finally de-bonded at the end of the treatment, with silicon impressions taken before adhesive removal.
  Other Names: Gemini metal brackets (3M Unitek)

SUMMARY:
Demineralisation and white-spot caries often occures during MB treatment. While resin infiltration has been proved to stop progression of enamel demineralisation, there is still a paucity of information in the literature concerning the best time point of infiltration: During or following MB treatment. Infiltration during treatment requires debonding respective brackets prior to infiltration, with subsequent re-bonding. In terms of preventing enamel damages by progression of demineralisation and enamel damages by de-bonding, it is unclear whether it was better to infiltrate enamel immediately, or to better postpone until completion of MB treatment.

This study thus aimes to evaluate if resin infiltration can prevent enamel damage due to bracket de-bonding.

DETAILED DESCRIPTION:
Background: Orthodontic bracket debonding is known to cause side-effects such as enamel cracks or fractures. There is a lack of information on potential benefits or side-effects of removing brackets from infiltrated enamel, in terms of enamel damages, in vivo.

Purpose: To assess enamel damages following debonding in demineralised teeth with or without prior infiltration (Icon, DMG, Hamburg, Germany), compared to those following bracket removal from sound enamel, in order to provide guidelines for the right time point of infiltration of post-orthodontic lesions (during or following orthodontic treatment).

Design: Single-center, randomized, single blinded, split-mouth controlled clinical trial Subjects: 30 subjects with fixed multi-bracket (MB) appliances treated at the orthodontic clinic of Dr. Roberto Vogel, Temuco, Chile: It is planned to include 20 consecutive patients with extensive decalcifications, and 10 patients without decalcifications. Random allocation of demineralized dental arch quadrants to the different treatment groups (debond with or without prior infiltration, and sound teeth).

Investigated tooth groups: Upper and lower canines, and upper and lower incisors.

Methods: Bracket bonding procedure (Transbond XT 3M, Unitek) is identical for all patients and also for the re-attachement of brackets. Teeth allocated to the infiltration group will receive bracket removal, infiltration and rebonding of new brackets 4 weeks prior to final debonding. De-bonding procedures are identical for all patients.

Silicone replicas are made directly following bracket removal (prior to adhesive removal). Replica analysis is performed using a confocal microscope (Zeiss LSM780) at the Department of Cell Biology, University of Concepción, Chile.

ELIGIBILITY:
Inclusion Criteria:

* Multibracket apparature with: At least 4 post-orthodontic white spots on front teeth (canines and / or incisors) in upper and lower jaw (study group) OR
* No post-orthodontic white spot or any other enamel damage - on front teeth (canines and / or incisors) in upper and lower jaw (control group) AND
* No cavitation of vestibular tooth surface(s) AND
* Patients willing to participate in the study and accepting to attend recall visits

Exclusion Criteria:

* Cavitation of vestibular tooth surface(s)
* Participation in other study
* History of allergy towards any dental material.
* Subjects with any systemic and local conditions not permitting the treatment
* Subjects with direct or indirect restorations in maxillary central or lateral incisors.
* Subjects not willing to participate in the study
* Subjects with fractured teeth maxillary central or lateral incisors
* No or less than 4 post-orthodontic white spots on front teeth (canines or incisors) in upper or lower jaw (study group)
* Post-orthodontic white spots or any other enamel damage on front teeth or incisors (control group)

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Surface damages | 4 weeks after deboning
  Number of cracks and fractures as assessed by enamel surface analysis via silicone replicas using CLSM

CONTACTS AND LOCATIONS:
Overall Officials: Michael Knösel, Principal Investigator — University Medical Center (UMG) Göttingen
Locations (1):
- Dental Clinic, Temuco, Región de la Araucanía, Chile